CLINICAL TRIAL: NCT03815253
Title: Electro-acupuncture for Central Obesity: a Single Blinded Randomized Sham-controlled Clinical Trial
Brief Title: Electro-acupuncture for Central Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Zhong Lidan, Research Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKBU-HMRF
Record Dates: First submitted 2019-01-12; First posted 2019-01-24 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Central Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: single-blinded, randomized, sham-controlled clinical trial
Who Masked: Participant
Masking Description: Subjects of both groups will be randomly assigned to receive either electro-acupuncture or control (sham) treatment. For randomization, simple, complete non-sequential random numbers will be generated in advance by a computer program in a block of four, and kept by the principal investigator. After a patient's eligibility is confirmed, a randomization number which corresponds to the group allocation will be provided to the acupuncturist by the PI. This arrangement will ensure that the clinical assessor and participants are blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Body electro-acupuncture will be conducted for 2 sessions per week over 8 consecutive weeks.
  Body electro-acupuncture will choose eight acupoints as Tianshu(ST-25), Daheng(SP-15), Daimai(GB-26), Qihai(CV-6), Zhongwan(CV-12), Zusanli (ST-36), Fenlong(ST-40), Sanyinjiao(SP-6).Disposable acupuncture needles (verum acupuncture needles asia-med Special No. 16 with 0.30 x 0.30mm matching the Streitberger sham-needles) will be inserted at a depth of 10-25 mm into the points.
  We will also deliver electrical stimulation with dense-disperse waves with 50Hz at 10 volts through electrical acupuncture stimulation instrument (ES-160 6-Channel Programmable Electro-acupuncture) to the abdominal points. The bodily needles will be retained for 30 minutes.
  Interventions: Other: acupuncture
- sham-acupuncture group (Placebo Comparator): As to the participants allocated to control group, Streitberger's non-invasive acupuncture needles (Gauge 8 x 1.2" / 0.30 x 30 mm) will be applied to act as sham control at the same acupoints with same stimulation modality. However, the needles will be only adhered to the skin instead of insertion. The validity and credibility of this model has been well demonstrated.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Body electro-acupuncture will choose eight acupoints as Tianshu(ST-25), Daheng(SP-15), Daimai(GB-26), Qihai(CV-6), Zhongwan(CV-12), Zusanli (ST-36), Fenlong(ST-40), Sanyinjiao(SP-6).Disposable acupuncture needles (verum acupuncture needles asia-med Special No. 16 with 0.30 x 0.30mm matching the Streitberger sham-needles) will be inserted at a depth of 10-25 mm into the points.
  We will also deliver electrical stimulation with dense-disperse waves with 50Hz at 10 volts through electrical acupuncture stimulation instrument (ES-160 6-Channel Programmable Electro-acupuncture) to the abdominal points. The bodily needles will be retained for 30 minutes.

SUMMARY:
In this study, a 8-week, single blinded, randomized controlled clinical trial will be conducted to examine the efficacy and safety of body acupuncture in the treatment of central obesity in Hong Kong.

DETAILED DESCRIPTION:
This is a pilot single-blind, randomized, sham-controlled trial. 168 central obesity patients will be randomly assigned to acupuncture group or control group. The duration of the treatment will be 8 weeks with 2 session per week and the follow-up period will be 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are defined as eligible participants: men and women aged between 18 and 65 years old; BMI ≥ 25 kg/m2; central obesity, defined as WC of ≥ 90 cm in men and ≥ 80 cm in non-pregnant women according to ICD-10 [24]; not receiving any other weight control measures or any medical and/or drug history in last 3months.

Exclusion Criteria:

Patients who meet any of the following criteria should be excluded from the study: endocrine diseases, including thyroid disorder, pituitary disorder, sex gland disorder, etc.; heart diseases, including arrhythmia, heart failure, myocardial infarction, patients with pacemaker; allergy and immunology diseases; bleeding tendency; pregnant or lactating women; impaired hepatic or renal function; stroke or unable to exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in waist circumference | 0,1,2,3,4,5,6,7,8, 11, 15,18, 21, 24 weeks
  Waist circumference will be measured around the abdomen at the level of the umbilicus (belly button).

SECONDARY OUTCOMES:
Changes in hip circumference | 0,1,2,3,4,5,6,7,8,9,11,15,18, 21, 24 weeks
  hip circumference measured at the level of maximum posterior extension of the buttocks
Adverse events after treatment and follow up | 0,1,2,3,4,5,6,7,8, 15,18, 21, 24 weeks
  Adverse events of acupuncture treatment will be assessed using the Treatment Emergent Symptom Scale (TESS) and would be evaluated during the whole procedure, as well as laboratory tests (whole blood counts, renal and liver functions) if needed. All clinical adverse events will be recorded in terms of intensity (mild, moderate, or severe), duration, outcome and relationship to the study.
Changes in waist-to-hip circumference ratio | 0,1,2,3,4,5,6,7,8, 15,18, 21, 24 weeks
  waist-to-hip ratio is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement ( W ÷ H ).
Changes in Body Mass Index | 0,1,2,3,4,5,6,7,8, 15,18, 21, 24 weeks
  Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Changes in body fat percentage | 0,1,2,3,4,5,6,7,8, 15,18, 21, 24 weeks
  The body fat percentage (BFP) of a human or other living being is the total mass of fat divided by total body mass, multiplied by 100. Body fat percentage will be measured by Omron Karada Scan HBF-701.
Changes in total cholesterol (TC), triglyceride (TG) and fasting blood glucose (FBG) | 0, 8 weeks
  Total cholesterol (TC), triglyceride (TG) and fasting blood glucose (FBG) will be measured before and after the 8-week treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxiang Bian, MD., Ph.D, Study Director — Hong Kong Chinese Medicine Clinical Study Centre
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lam TF, Lyu Z, Wu X, Wong YP, Cao P, Wong EY, Hung HB, Zhang S, Bian Z, Zhong LLD. Electro-acupuncture for central obesity: a patient-assessor blinded, randomized sham-controlled clinical trial. BMC Complement Med Ther. 2024 Jan 29;24(1):62. doi: 10.1186/s12906-024-04340-5. PMID 38287303
- [Derived] Zhong LLD, Wu X, Lam TF, Wong YP, Cao P, Wong EY, Zhang S, Bian Z. Electro-acupuncture for central obesity: randomized, patient-assessor blinded, sham-controlled clinical trial protocol. BMC Complement Med Ther. 2021 Jul 3;21(1):190. doi: 10.1186/s12906-021-03367-2. PMID 34217283